CLINICAL TRIAL: NCT01274143
Title: Impact of Remote Familial Colorectal Cancer Assessment and Counseling
Brief Title: Family Colorectal Cancer Awareness and Risk Education Project (Family CARE Project)
Acronym: Family CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Anita Kinney, Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB_00017894; 7R01CA125194-06 (NIH)
Record Dates: First submitted 2010-12-10; First posted 2011-01-11 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2015-05

CONDITIONS: Colorectal Cancer
Keywords: Colorectal; Cancer; Colon; Rectal; Behavioral Intervention; Screening; Motivational Interviewing; Extended Parallel Process Model; Implementation Intentions; Family CARE
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telephone-delivered risk intervention (Active Comparator): Participants in this arm receive a personalized telephone-risk assessment intervention provided by a trained cancer risk counselor.
  Interventions: Behavioral: TeleCARE
- Mailed pamphlet intervention group (Active Comparator): Participants in this group receive a mailed pamphlet containing information about familial colorectal cancer risk and screening.
  Interventions: Behavioral: Pamphlet intervention

INTERVENTIONS:
Behavioral: TeleCARE — Personalized telephone-delivered cancer risk assessment.
  Arms: Telephone-delivered risk intervention
Behavioral: Pamphlet intervention — Mailed pamphlet about familial colorectal cancer risk and screening.
  Arms: Mailed pamphlet intervention group

SUMMARY:
The Family Colorectal Cancer Awareness and Risk Education Project (Family CARE Project) is designed to determine whether a personalized telephone plus mailed print cancer risk assessment and behavior change counseling intervention is more effective than a targeted mailed print intervention in promoting risk appropriate screening in individuals with a family history of the disease. The project targets people residing in both rural and urban areas, allowing an examination of differential intervention effects with regard to place of residence.

DETAILED DESCRIPTION:
The rate of adherence to regular colonoscopy screening (CS) among members of families at increased risk for colorectal cancer (CRC) is far below recommended levels. Persons who live in rural areas of the United States exhibit lower CRC screening rates than their urban counterparts. Although the detection of familial predisposition to cancer begins with an accurate family medical history, data indicate that many patients do not receive adequate familial cancer risk assessment from their primary care providers. This suggests that familial risk is largely unrecognized which may lead to inadequate risk stratification, lack of risk notification, appropriate risk counseling, suboptimal cancer screening and preventable deaths. Because of geographic and system-level barriers, special efforts are needed to improve access to personalized risk communication and adherence to CRC screening to rural and other geographically underserved populations at increased risk for CRC. In the proposed study, we will evaluate a novel telephone-based, theory-guided personalized risk communication intervention that combines a familial CRC risk assessment and behavioral counseling with tailored messages. The key hypothesis guiding this study is that a multifaceted personalized risk communication intervention will improve CS at a significantly higher rate than a mailed targeted print intervention.

Our integrative study model specifies important theoretical mechanisms that can contribute to increased use of CS among persons at increased risk. We will enroll 438 adult men and women between the ages of 30-74 who are considered at increased risk of familial CRC into this 2-group randomized trial. The primary aim of this study is to compare colonoscopy use among participants in the two groups. Secondary aims are to compare the two groups with regard to cognitive and emotional outcomes and explore the underlying mechanisms through which the interventions have an impact on colonoscopy behavior. Sociodemographic, clinical, behavioral and psychosocial measures will be collected from participants at baseline, and 1 month, 9 months, and 15 months following the intervention. Self-reported colonoscopy is verified with medical records.

The study's findings will have both theoretical, as well as practical significance. Our findings will help to influence the selection and dissemination of effective outreach approaches to improve CRC screening in populations at increased risk for the disease. These results have broad applicability to understanding responses to personalized risk communication interventions for other diseases as well. Findings will also broaden our understanding of the underlying theoretical mechanisms of how remote cancer risk communications lead to improvements in cancer screening among geographically underserved populations if such intervention effects are observed.

In addition to studying the intervention effects in rural areas, we will enroll participants in urban areas. These enhancements to our population-based randomized behavioral trial will provide us with an unprecedented opportunity to assess reach and determine if there are differential intervention effects (i.e., efficacy) with regard to place of residence (rurality vs. urbanicity.)

ELIGIBILITY:
Inclusion Criteria:

* Have at least one first-degree relative diagnosed with colorectal cancer (CRC) between the ages of 40-59, or one first-degree relative diagnosed with colorectal cancer at age 40 or older and an additional first-degree or second-degree relative diagnosed with colorectal cancer at age 40 or older.
* If relative was diagnosed over age 50, participant must be 40-74 years old.
* If relative was diagnosed at age 40-49, participant cannot be more than ten years younger than relative at first diagnosis (e.g., dx at 48, participant must be 38-74 years old).
* Colorectal cancer cases of relatives recruited through the cancer registries of California, Colorado, Idaho, New Mexico, or Utah; Rocky Mountain Cancer Genetics Coalition sites of National Cancer Genetics Network in Colorado, New Mexico, or Utah; or Intermountain Health Care

Exclusion Criteria:

* Previous cancer diagnosis of any kind (except for non-melanoma skin cancers).
* Has had a colonoscopy within the past five years.
* Meets clinical criteria for Lynch syndrome or other polyposis syndromes.
* Has had prior involvement in colorectal cancer-related clinical, behavioral or epidemiologic cancer familial research.
* Mentally incompetent, incarcerated, hearing or visually impaired.
* Unable to read and speak English fluently.

Ages: 30 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2008-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Colonoscopy | 9 month follow-up
  The primary outcome is colonoscopy. Medical record verification of self-reported colonoscopy is performed.

SECONDARY OUTCOMES:
Fecal occult blood test (FOBT)/Fecal Immunochemical Test (FIT) | Baseline, 1 month, 9 month, and 15 month follow-up
  Fecal occult blood test(FOBT) following the intervention. Medical confirmation of self-reported FOBT/FIT is performed.
Perceived Control | Baseline, 1 month and 9 month follow-up
  The Perceived Personal Control Scale is an integrative outcome that encompasses the broad spectrum of health risk communication and informed decision-making. This validated scale is a 9-item measure representing three dimensions of control participants believe they have regarding family history of colorectal cancer (CRC): cognitive-interpretive, decisional, and behavioral. A 5-point Likert-style response format is used ranging from very little control to very high control. A total scale score is calculated by summing the items.
Perceived Risk | Baseline, 1 month and 9 month follow-up
  A 4-item scale with established construct and predictive validity with regard to cancer screening will assess participants' subjective perceived risk for developing colorectal cancer. Responses are measured on a five-point Likert scale ranging from very small to very large.
Psychological distress | Baseline, 1 month and 9 month follow-up
  Generalized psychological distress will be operationalized as state anxiety and we will use the State Subscale of the State Trait Anxiety Inventory. We will also measure cancer-specific distress with the Impact of Event Scale. The stressor in this study is having a family history of colorectal cancer.
Knowledge | Baseline, 1 month and 9 month follow-up
  The Colorectal Cancer Knowledge Survey is a validated 12-item scale that assesses colorectal cancer screening knowledge, colorectal cancer risk factors (including family history) and CRC symptoms. The questionnaire consists of true/false with a possible range of scores of 0-12. FOBT items will be substituted with colonoscopy.
Decisional Conflict | Baseline, 1 month and 9 month follow-up
  Participants are asked to evaluate whether or not they feel confident in their decision to receive or not receive CRC screening. Assessment following the intervention will determine whether the decisional conflict has been resolved and whether or not that resolution results in colonoscopy uptake.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Y Kinney, Ph.D., R.N., Principal Investigator — Huntsman Cancer Institute and University of Utah
Locations (8):
- United States (8):
  - California Cancer Registry, Sacramento, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Colorado Central Cancer Registry, Denver, Colorado
  - Cancer Data Registry of Idaho, Boise, Idaho
  - University of New Mexico, Albuquerque, New Mexico
  - Intermountain Health Care, Salt Lake City, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Utah Cancer Registry, Salt Lake City, Utah

REFERENCES:
- [Derived] Brumbach BH, Birmingham WC, Boonyasiriwat W, Walters S, Kinney AY. Intervention Mediators in a Randomized Controlled Trial to Increase Colonoscopy Uptake Among Individuals at Increased Risk of Familial Colorectal Cancer. Ann Behav Med. 2017 Oct;51(5):694-706. doi: 10.1007/s12160-017-9893-1. PMID 28236077
- [Derived] Anderson AE, Flores KG, Boonyasiriwat W, Gammon A, Kohlmann W, Birmingham WC, Schwartz MD, Samadder J, Boucher K, Kinney AY. Interest and informational preferences regarding genomic testing for modest increases in colorectal cancer risk. Public Health Genomics. 2014;17(1):48-60. doi: 10.1159/000356567. Epub 2014 Jan 14. PMID 24435063
- [Derived] Boonyasiriwat W, Hung M, Hon SD, Tang P, Pappas LM, Burt RW, Schwartz MD, Stroup AM, Kinney AY. Intention to undergo colonoscopy screening among relatives of colorectal cancer cases: a theory-based model. Ann Behav Med. 2014 Jun;47(3):280-91. doi: 10.1007/s12160-013-9562-y. PMID 24307472
- [Derived] Simmons RG, Lee YC, Stroup AM, Edwards SL, Rogers A, Johnson C, Wiggins CL, Hill DA, Cress RD, Lowery J, Walters ST, Jasperson K, Higginbotham JC, Williams MS, Burt RW, Schwartz MD, Kinney AY. Examining the challenges of family recruitment to behavioral intervention trials: factors associated with participation and enrollment in a multi-state colonoscopy intervention trial. Trials. 2013 Apr 30;14:116. doi: 10.1186/1745-6215-14-116. PMID 23782890